CLINICAL TRIAL: NCT05901194
Title: Study of the Benefit of Lenvatinib Treatment in Waiting List of Liver Transplantation After TACE Failure in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Lenvatinib Treatment in Waiting List of Liver Transplantation After TACE Failure in Patients With Hepatocellular Carcinoma
Acronym: Ta-Len-Tra
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoire EISAI (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP220267; 2022-000998-31 (EudraCT Number)
Record Dates: First submitted 2023-05-26; First posted 2023-06-13 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Liver transplantation; non resectable hepatocellular carcinoma
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib (Experimental): Lenvatinib will be administred orally and daily at the usual dose ( 8 or 12 mg per day depending on the weight < or ≥ 60kg) in the 25 patients of the study from TACE failure until LT
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administred orally and daily at the usual dose ( 8 or 12 mg per day depending on the weight < or ≥ 60kg) in the 25 patients of the study from TACE failure until LT

SUMMARY:
Currently in France, hepatocellular carcinoma (HCC) represents over 30% of indications of liver transplantation (LT) (# 500 cases/year). Chemoembolization (TACE) is the most commonly used bridge treatment in those patients (estimate 60%). These patients will present with a complete response in only 60 % of the cases (# 180 patients per year in France) and failure in 40 % of the cases (# 120 patients per year in France).

A systemic treatment using lenvatinib might provide a benefit in patients presenting with a non-resectable HCC in waiting list for LT and with a TACE failure (i.e. those with an active disease and a partial response or a stable disease or a progressive disease on imaging data, in particular when AFP remains significantly increased after 2 TACE) by decreasing dropout rate before LT and decreasing recurrence rate post-LT without new safety signal.

DETAILED DESCRIPTION:
The investigators identified a sub-group of patients with non resectable HCC that could benefit from a systemic neoadjuvant medical strategy before liver transplantation (LT). In these patients, the investigators propose to add oral systemic chemotherapy with lenvatinib as a bridging/downstaging therapeutic approach until LT.

In the case of at least partial response or stability under lenvatinib and within AFP score of 2, the patients will be transplanted and lenvatinib will be stopped on the day or the day before LT (depending on the availability of the graft).

In the case of disease progression, the patient will stop prematurely the lenvatinib treatment and will be treated according to usual practices. The patient's eligibility for LT will be assessed according to usual practices.

ELIGIBILITY:
Inclusion Criteria:

* Non resectable HCC
* Initial French AFP score < or = 2
* Registered on national waiting list for LT
* Who underwent TACE as a bridge to LT
* With no complete response after 2 TACE (i.e. persistent active disease, including stable disease or partial response or progression)
* Non eligible for percutaneous ablation
* Informed, written consent obtained from the patient
* Having the rights to French social insurance
* Aged of 18 years or older
* Adequate bone marrow, liver and renal function as assessed by the following laboratory tests:

  * Hemoglobin > 8.5 g/dL
  * Absolute neutrophil count ≥ 1500/mm3 (≥ 1200/mm3 for black/African, American)
  * Platelet count ≥ 60,000/ mm3
  * Total bilirubin ≤ 2 mg/dL or 34 mcmol/l
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN)
  * Serum creatinine ≤ 1.5 x ULN
  * Prothrombine time-international normalized ratio (PT-INR) < 2.3 and PTT < 50 %
  * Glomerular Filtration Rate (GFR) ≥ 30 mL/min/1.73 m2
* Patient with QT/QTc < 480 ms
* Women of childbearing potential (WOCBP) need to accept one effective method of contraception until 1 month after the last lenvatinib intake and avoid pregnancy
* Patients who are sexually active with WOCBP partners need to accept one effective method of contraception until 1 month after lenvatinib intake and men must agree to use adequate contraception.

Exclusion Criteria:

* Contraindication of lenvatinib and excipient

  1. Cardiovascular:

     * Rhythmic or ischemic recent or uncontrolled cardiac disease: Pacemakers or patients who have a history of cardiac arrhythmias or irregular heartbeats (in case of electroporation procedure)
     * Congestive heart failure New York Heart Association (NYHA) ≥ class 2
     * Unstable angina or myocardial infarction within the past 6 months before enrolment
     * Uncontrolled arterial hypertension (systolic ≥ 140 mmHg, diastolic ≥ 90 mmHg)
  2. Ongoing ascites: Refractory ascites according to EASL guidelines definition (ascites that cannot be mobilized or the early recurrence of which cannot be prevented because of a lack of response to sodium restriction and diuretic treatment)
  3. Coagulopathy
  4. Ongoing infection > Grade 2 according to NCI-current CTCAE . Hepatitis B is allowed if no active replication is present (below 100 IU/mL). Hepatitis C is allowed if no antiviral treatment is ongoing
* Known hypersensitivity to the study drug or excipients in the formulation
* Decompensated cirrhosis (Child-Pugh > A6)
* Prior systemic therapy with oral TKI and/or immunotherapy
* Past or concurrent history of neoplasm other than HCC, except for in situ carcinoma of the cervix uteri and/or non-melanoma skin cancer and superficial bladder tumours. Any cancer curatively treated > 3 years prior to study entry is permitted
* Recent digestive bleeding associated with portal hypertension (whithin the 3 months prior to inclusion in the study)
* Advanced or Metastatic HCC (BCLC C)
* Persistent proteinuria of NCI-current CTCAE ≥ Grade ≥ Grade 3
* Project of living donor
* Pregnant or lactating woman
* Curator or guardianship or patient placed under judicial protection
* Participation in other interventional research during the study.
* History within the past 3 months before enrollment of haemorrhage, gastrointestinal perforation, gastrointestinal or non-gastrointestinal fistula,
* History of aneurism,
* Hypokalemia, hypomagnesemia and hypocalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with lenvatinib who have a Liver transplantation (LT) | 12 months
  The proportion of patients with TACE failure and treated with lenvatinib who have a LT

SECONDARY OUTCOMES:
Time to progression under lenvatinib | up to 12 months and until LT
  Time to progression under lenvatinib before LT by imaging. Progression will be based on RECIST and mRECIST
Progression under lenvatinib | up to 12 months and until LT
  Progression under lenvatinib before LT by imaging. Progression will be bases on RECIST and mRECIST
Response rate | up to 12 months and until LT
  Response rate before LT by imaging
Response rate | after the LT, during 18 months
  Response rate by liver specimen pathology after the LT
Recurrence rate | after LT, during 18 months
  Recurrence rate after LT by imaging
Incidence of Treatment-Emergent Adverse Events | Throughout the study, an average of 31 months
  Incidence of Treatment-Emergent Adverse Events using current CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ROSMORDUC, Principal Investigator — APHP, Paul Brousse Hospital, villejuif, France
Locations (6):
- France (6):
  - Hospital Haut levêque, Bordeaux
  - Hospital Henri Mondor, Créteil
  - Hospital Claude Huriez, Lille
  - Pontchaillou Hospital, Rennes
  - Hospital Trousseau, Tours
  - Paul Brousse Hospital, Villejuif

IPD SHARING:
Plan to Share IPD: No